CLINICAL TRIAL: NCT02470442
Title: Sevoflurane Vs. Sevoflurane-desflurane Anesthesia in Children With Laryngeal Mask Airways; Difference in Respiratory Event, Recovery Time and Emergence Agitation
Brief Title: Desflurane in Children With Laryngeal Mask Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-1504-116-668
Record Dates: First submitted 2015-06-08; First posted 2015-06-12 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Desflurane Anesthesia
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane/Desflurane (Experimental): After induction of general anesthesia with sevoflurane, anesthesia was maintained with desflurane.
  Interventions: Drug: Sevoflurane/Desflurane
- Sevoflurane (Experimental): the anesthetic induction and maintenance with sevoflurane.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane/Desflurane — Anesthesia induced with sevoflurane and anesthetic maintenance with desflurane
  Other Names: suprane
  Arms: Sevoflurane/Desflurane
Drug: Sevoflurane — Anesthesia induced with sevoflurane and anesthetic maintenance with sevoflurane
  Arms: Sevoflurane

SUMMARY:
The purpose of this study is to characterize the airway responses to desflurane during maintenance of and emergence from anesthesia in children whose airways were supported with laryngeal mask airways (LMAs).

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective surgery under general anesthesia with laryngeal mask airway

Exclusion Criteria:

* history of reactive airways disease with an acute exacerbation within the past 2 weeks
* if wheezing or an active upper respiratory infection was present on the day of surgery
* if there was a history of malignant hyperthermia
* a history of moderate-to-severe hepatic dysfunction following anesthesia with desflurane not otherwise explained.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
respiratory adverse events | participants will be followed for postoperative period, an expected average of 30 minutes.

SECONDARY OUTCOMES:
emergence agitation | 15 minutes after arrival on PACU

CONTACTS AND LOCATIONS:
Overall Officials: JinTae Kim, MD. PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea